CLINICAL TRIAL: NCT01630525
Title: " The Eyes Have it " : Ocular Saccade Abnormalities in Prodromal Alzheimer's Disease
Acronym: LYLO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2011/22
Record Dates: First submitted 2012-06-21; First posted 2012-06-28 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; neurodegenerative signs
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Prodromal AD participants
  Interventions: Other: Neuropsychological assessment; Other: ophthalmologic checkup; Other: Automated non-invasive oculometry
- Typical AD participants
  Interventions: Other: Neuropsychological assessment; Other: ophthalmologic checkup; Other: Automated non-invasive oculometry
- Control participants
  Interventions: Other: Neuropsychological assessment; Other: ophthalmologic checkup; Other: Automated non-invasive oculometry

INTERVENTIONS:
Other: Neuropsychological assessment — Neuropsychological assessment : MMSE (Greco), RL/RI-16 items (Van der Linden 2003), visual retention test (DMS48), verbal fluency (Thurstone et Thurstone 1964), TMT A and B (Reitan 1956), DSST (Weschler 1997), Clinical Dementia Rating Scale (Hughes 1982), image naming DO80 (Deloche et Hannequin 1997), Similarities and Digit Span subscores of the WAIS (Weschler 1997), Anxiety and Depression (GDS), activities of daily living (ADL-Katz and IADL-Lawton).
Other: ophthalmologic checkup — Vision work-up, 30 minutes (VA, non invasive retinal imaging : non dilated optic fundus picture or OCT, ocular tension).
Other: Automated non-invasive oculometry — Automated non-invasive oculometry : 45 minutes with rest periods : horizontal and vertical pro- and anti-saccades, prediction, spatial decision (Monsiman et al. Brain 2005,128:1267-127, items detection (Rösler et al. Cortex 2005 ;41 :512-519) and exploration/curiosity of non congruent images and faces according to Daffner et al. Neurology 1992 ;42 :320-328 and Loughland et al. Biol Psychiatry 2002 ;52 : 338-348).

SUMMARY:
Alzheimer's disease (AD) has a prolonged prodromal phase before the stage of dementia. Subtle executive cognitive function deficits can be detected at this early pre-dementia phase, more than 10 years before dementia. Among them, the digit symbol substitution task (DSST) has been shown to be altered very early, up to 13 years before dementia. This test, as many others executive function tests, requires a fine control of visuomotor coordination. Like executive functions, eye movements, particularly voluntary-guided saccades, are under the control of the frontal lobe and fronto-parietal networks. Previous studies have shown a deterioration of voluntary saccades in AD using various paradigms. There are no data in prodromal AD, although the pathological process of the disease affects very early brain structures implicated in saccades execution (eg. caudate nucleus and pre-cuneus).

ELIGIBILITY:
Inclusion Criteria:

All patient groups:

* Age >60 years
* Normal vision work-up : (corrected binocular visual acuity > 8/10)
* Written informed consent
* Subjects affiliated to Social Security

Group A: Prodromal AD.

* Memory complaints.
* Normal or slight restriction of IADL.
* "hippocampal-type" amnesic syndrome defined by poor free recall despite adequate (and controlled) encoding, decreased total recall because of insufficient effect of cuing or impaired recognition, numerous intrusions (RL/RI-16items)
* CDR (Clinical Dementia Rating Scale) ≥ 0,5
* Persistence of memory changes at a subsequent assessment (>3 months)
* Absence of global cognitive deterioration (MMSE ≥24)
* Exclusion of other disorders that may cause mild cognitive impairment with adequate tests
* 1.5 Tesla diagnosis MRI with at least T2, Flair transversal sections and coronal T1 sections in the coronal plan. Absent or slight medio temporal/hippocampal atrophy or if available (non mandatory) characteristic CSF betaA42/tau ratio

Group B: Typical AD (mild to moderate)

* NINDS-ADRDA diagnosis criteria
* MMSE ≥ 20

Group C: Control subjects

* No memory or other significant cognitive complain.
* MMSE ≥ 24

Exclusion Criteria:

All groups :

* Clinically significant vision abnormality(P8 without glasses)
* Oculomotor deficit or strabismus
* Depression (GDS) with treatment
* Subjects unable to give their informed consent

Controls :

* Memory or any other significant cognitive complain.
* Abnormalities at inclusion (V0) neuropsychology testing suggestive of a cognitive deficit.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A : 30 Prodromal Alzheimer Disease, Group B : 30 typical Alzheimer Disease, Group C : 30 controls age-matched ± 5 years to Group A (to Group A) Total of 90 subjects.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Saccades execution parameters | Study visit (Up to 1 month after inclusion)
  To demonstrate the alteration of saccade execution parameters (latency, velocity, precision, errors) during pro and anti-saccades, spatial decision and prediction tasks in prodromal AD compared to mild to moderate AD and aged-matched controls.
  Variables recorded :
  Saccades execution parameters :
  * Mean latency (msec),
  * Mean velocity (°/msec) and maximal velocity,
  * Accuracy or mean gain,
  * Mean percent of errors and corrected errors,
  * Mean percent of prediction.

SECONDARY OUTCOMES:
Neuropsychology tests scores | At inclusion (Day 0)
Pre-defined variables on visual exploration tasks (fixation number and durations, errors). | Study visit (Up to 1 month after inclusion)
Number of point fixation in degraded areas and of visual attention induced cards | Study visit (Up to 1 month after inclusion)

CONTACTS AND LOCATIONS:
Overall Officials: François TISON, Pr, Principal Investigator — University Hospital, Bordeaux; Geneviève CHENE, Pr, Study Chair — University Hospital, Bordeaux
Locations (3):
- France (3):
  - Lyon UniversityHospital, Lyon
  - AP-HM, Marseille
  - CHU de Bordeaux Hôpital Haut Lévêque, Pessac